CLINICAL TRIAL: NCT03404999
Title: Automated Clinical-Decision Support to Improve Hypertension Care Among Overweight Children in Primary Care
Brief Title: Clinical-Decision Support to Improve Hypertension Care in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STU 052015-029
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Blood Pressure; Overweight and Obesity
MeSH Terms: conditions — Hypertension; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Four-month time series trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- clinical decision support activated (Experimental): TWO MED ASSIST ALERTS
  1. Enter height (when missing)
  2. Repeat BP (when high)
  ONE PROVIDER ALERT
  1. BP high & prior BP/BP%s
  2. Defines elev. BP, HTN stage 1-2 with button to enter diagnosis
  3. Link to tailored ordersets
  TAILORED ORDERSETS
  1. Elevated BP
     1. Button to schedule f-up <6 m
     2. Button for diet/lifestyle counseling/check-out instructions
  2. HTN stage 1
     1. Buttons to order labs/studies pre-checked for stage 1 recs
     2. Button for nephrology referral
     3. Button to schedule f-up in 1-2 wk/<1 m
     4. Button for diet/lifestyle counseling/check-out instructions
  3. HTN stage 2
     1. Buttons to order labs/studies for stage 2
     2. Button for nephrology referral (pre-checked)
     3. Button to f-up 1 wk
     4. Button for diet/lifestyle counseling/check-out instruction
  Interventions: Other: clinical decision support

INTERVENTIONS:
Other: clinical decision support — Decision support system (see description of hypertension decision support system alerts and order sets for details)

SUMMARY:
Approaches are needed to help primary-care pediatricians address high blood pressure. This study will test whether an electronic health-record-based tool to address high blood pressure is feasible and improves the evaluation and management of high blood pressure in clinical practice. If successful, this approach can be used to address other lifestyle-related and complex health problems (e.g., dyslipidemia and diabetes), then disseminated and used nationwide.

The investigators have developed a new, electronic health-record (EHR)-based tool that is designed to help pediatricians:

1. IDENTIFY AND DOCUMENT

   1. when a child's blood pressure is elevated, and
   2. whether it has been elevated before--including number of prior elevations to document the correct diagnosis (for example, elevated blood pressure, vs. hypertension stage 1, vs. hypertension stage 2), THEN
2. ORDER the next action(s) needed per guideline-based recommendations, AND per prior actions taken--including:

   1. laboratories and studies per 2017 updated guidelines
   2. follow-up interval in primary care
   3. referral to nephrology, when indicated, and
   4. patient education on diet/lifestyle modification.

The investigators are working on improving this system further with addition of orders for:

1. referral for sleep-apnea testing and treatment, when indicated, and
2. blood-pressure medications (for example, initiation, titration, or addition of agents depending on blood-pressure control, comorbid conditions [e.g., diabetes], and risk for pregnancy)

DETAILED DESCRIPTION:
The investigators' data suggest that (1) addressing obesity-related comorbidities (in combination with high BMI/overweight/obesity) and more frequent follow-up are associated with weight-status improvement in overweight (OW) children, (2) that parents rank checking for weight-related health problems as the #1 most important recommended weight-management clinical practice, but that (3) comorbidities are infrequently addressed. Thus, to improve weight status, interventions are needed to improve comorbidity identification, evaluation, and management in primary care. Because the investigators' data suggest that identification of high blood pressure is particularly poor, and that identifying blood-pressure elevations in young children at three separate encounters is complex, they are using existing underutilized data to automate addressing high blood pressure/hypertension in an electronic health record system (EPIC-based), and, if successful, applying the method to other obesity-related comorbidities in primary care.

OF NOTE: in developing and pilot-testing this decision support tool, providers wanted access to it for patients without overweight/obesity. Thus, although the trial was borne out of work in weight-management research, the initial trial will focus on all children irrespective of weight status.

ELIGIBILITY:
Inclusion Criteria for Providers: Pediatric primary care providers practicing at participating clinics that have agreed to have the decision-support system implemented.

Exclusion Criteria for Providers:

* Lack of electronic health record

Inclusion Criteria for Children:

* Measured systolic or diastolic blood pressure >=90th % for age/sex, or
* >=120 mmHg systolic or >=80 mmHg diastolic (whichever is lower)

Exclusion Criteria for Children:

* Diagnosis/visit for high blood pressure or hypertension in past 2 years
* Taking anti-hypertensive medication

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2803 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
High blood pressure addressed | 4-month time series analysis
  Proportion of patients with high blood pressure addressed post decision-support implementation (vs. pre-), defined as proportion of patients with elevated blood pressures or higher who have one or more diagnosis or orders placed to diagnose, evaluate, or manage hypertension. We will compare the slope of the post- vs. pre-implementation periods to examine change in monthly rate of HTN eval/management (indicated elements ordered/patients eligible) related to decision support that are in excess of secular trends in clinical practice. In the post-implementation period, the denominator will be determined by tracking patient-level decision-support fires. In the pre-implementation period, the denominator will be determined by applying the decision-support algorithm to retrospective data in monthly increments to identify patients who would have been eligible.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Parkland Medical Center, and (pilot took place at Children's Health), Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data are being obtained under a MU agreement/legal contract